CLINICAL TRIAL: NCT05777616
Title: The Impact of Medication Belief on Adherence to Infliximab in Patients With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0592
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's disease; adherence; medication concern; infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The IFX adherence to CD in China was not high. Medicine concerns may be predictive factor of adherence. By enhancing knowledge and relieving medicine concerns, we may increase patients' adherence to IFX.

DETAILED DESCRIPTION:
Crohn's disease (CD) is an incurable chronic disease that requires long-term treatment. As an anti-tumor necrosis factor (TNF) agent, Infliximab (IFX) is widely used in the treatment of Crohn's disease, while the adherence is not high. The purpose of this study was to investigate the adherence to IFX among CD patients in China and evaluate the association between medication belief and IFX adherence.

ELIGIBILITY:
Inclusion Criteria:

* patients with a confirmed diagnosis of CD; were treated with infliximab for at least 12 weeks; were informed consent.

Exclusion Criteria:

* The exclusion criteria were received treatment from mental health professionals due to any mental or cognitive impairment; suffered from other serious diseases, such as heart, brain, lung, liver and kidney dysfunction; severe infection, anemia, cachexia or other serious complications were found.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was conducted at the Second Affiliated Hospital, Zhejiang University School of Medicine (SAHZU) from November 15 to December 28, 2021. All CD patients treated with infliximab were retrospectively identified in the electronic medical records (EMRs) from the SAHZU Crohn's and Colitis Center.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Adherence | November 15 to December 28, 2021
  Adherence was judged by comparing the theoretical infusion times with the actual infusion times in recent 1 year, which was referred to the definition of modified medication possession radio (mMPR)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University,China
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China, Zhejiang, China